CLINICAL TRIAL: NCT05331339
Title: Effectiveness in Real Life of the Insulia® Digital Tool in Patients with Type 2 Diabetes Treated with Basal Insulin Therapy As Part of a National Telemedicine Program (ETAPES)
Brief Title: Real-life Efficacy of Insulia® Tool in Patients Living with Type 2 Diabetes Treated with Basal Insulin Therapy As Part of a National Telemedicine Program (ETAPES)
Acronym: INSULIA
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Sud Francilien (Other)
Responsible Party: Sponsor
Other Study IDs: 2022/0004
Record Dates: First submitted 2022-04-08; First posted 2022-04-15 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this study was to evaluate the INSULIA digital tool (automation of basal insulin dose calculation in type 2 diabetes) within the framework of a French national telemedicine experimentation program (ETAPES) in a single-center study.

The assumption is that a better metabolic control with this tool.

DETAILED DESCRIPTION:
Basal insulin titration in people with type 2 diabetes is of major importance to obtain the optimal dose to regulate fasting blood glucose without hypoglycemia.

Significant inertia in treatment optimization has been observed among both general practitioners and diabetologists.

The INSULIA tool (automation of basal insulin dose calculation in type 2 diabetes) within the framework of a French national telemedicine experimentation program (ETAPES) has been supported by the health authorities.

The data collected are of a single-center cohort of adult patients with type 2 diabetes who used this tool between 2018 and 2021.

It is supposed that a better metabolic control with this tool and aimed to understand factors associated with better results.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old.
* Patients with type 2 diabetes.
* Initiation or adjustment of basal insulin.
* Prescription of Insulia® for more than 6 months (between august 2018 and june 2021)
* Informed patient not opposed to the research

Exclusion Criteria:

Patient opposed to the research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Single-center diabetes department of a French public hospital.
Sampling Method: Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2022-11-02 (Actual); Primary Completion 2022-12-02 (Actual); Study Completion 2022-12-02 (Actual)

PRIMARY OUTCOMES:
HbA1c | at 6 months
  Evolution of HbA1c between baseline and 6 months after Insulia initiation

SECONDARY OUTCOMES:
Insulin | at 6 months
  Evolution of daily dose of basal insulin between baseline and 6 months after Insulia initiation
HbA1c objective | at 6 months
  Percentage of patients reaching the HbA1c target after 6 months
Mean fasting glucose | at 6 months
  Percentage of patients reaching a mean fasting glucose < 150 mg/dL for 7 days after 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Sud Francilien, Corbeil-Essonnes, France